CLINICAL TRIAL: NCT02378519
Title: Individualised Interactive Web-based Self-help Program and CBT-coaching in Combination With Physiotherapy for Patients With Persistent Musculoskeletal Pain
Brief Title: Interactive Web-based Program and CBT-coaching With Physiotherapy for Patients With Chronic Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luleå Tekniska Universitet (Other)
Collaborators: County Council of Norrbotten, Sweden (Other Government)
Responsible Party: Principal Investigator, Peter Michaelson, Senior lecturer, Luleå Tekniska Universitet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHSAM3_TAILORED_WEB_SSED
Record Dates: First submitted 2014-09-10; First posted 2015-03-04 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Musculoskeletal Pain
Keywords: Low back pain,; neck pain,; chronic pain; SSED; Pilot project; interactive web-based self-help programme; CBT-coaching; physiotherapy
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain; Neck Pain; Chronic Pain | interventions — Alkalies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-prog, followed by CBT + PT (Experimental): This arm of the single system experimental design starts with a baseline phase of 8 weeks where the subjects are introduced into to the interactive web-based self-help program. The baseline-period is followed by the intervention period which consists of a continued use of the interactive web-based self-help program, now with with cognitive behavioral therapy coaching in combination with individually tailored physiotherapy according to the person's needs for 16 weeks.
  Interventions: Behavioral: Base, followed by Web + CBT + PT
- Base, followed by Web + CBT + PT (Active Comparator): The intervention consists of a interactive web-based selfadministrated program with cognitive behavioral therapy coaching in combination with tailored physiotherapy according to the person's needs for 16 weeks.
  Interventions: Behavioral: Web-prog, followed by CBT + PT

INTERVENTIONS:
Behavioral: Web-prog, followed by CBT + PT — This arm of the single system experimental design starts with a baseline phase of 8 weeks where the subjects are introduced into to the interactive web-based self-help program. The baseline-period is followed by the intervention period which consists of a continued use of the interactive web-based self-help program, now with with cognitive behavioral therapy coaching in combination with individually tailored physiotherapy according to the person's needs for 16 weeks.
  Arms: Base, followed by Web + CBT + PT
Behavioral: Base, followed by Web + CBT + PT — The intervention consists of a interactive web-based selfadministrated program with cognitive behavioral therapy coaching in combination with tailored physiotherapy according to the person's needs for 16 weeks.
  Arms: Web-prog, followed by CBT + PT

SUMMARY:
The aim of the study is to evaluate the effects of a the multimodal treatment with a web-based self-help program with cognitive behavioral therapy coaching and individual tailored physiotherapy on workability, health behavior and pain symptoms for persons with persistent pain.

DETAILED DESCRIPTION:
Purpose The aim of the study is to evaluate the effects of a the multimodal treatment with a web-based self-help program with cognitive behavioral therapy (CBT) coaching and individual tailored physiotherapy on workability, health behavior and pain symptoms for persons with persistent pain.

Design In this study, we will apply a Single Subject Experimental Design (SSED) with a six week baseline phase, a 16 week intervention phase and a six week follow-up phase after twelve month. Outcome measurements will be performed regularly during all phases.

Participants Approximately 12 participants, fulfilling inclusion and exclusion criteria will be included in the study.

Inclusion criteria:

Persons, with persistent or recurrent pain from the neck-shoulder or back, with a duration for at least three months, aged 18-63 years, scoring ≥ 90 on Linton´s questionnaire, indicating risk for continuous sick leave and development of persistent pain, who are disposable for labor market at least 25% are eligible for the study. The participants have to be fluent in the Swedish language.

Exclusion criteria:

Patients with dementia and/or restricted cognitive functioning. Persons with depression and/or anxiety. The latter will be screened with the Hospital Anxiety Depression Scale questionnaire. Terminally ill patients, comorbidity which might prevent treatment participation and ongoing causal treatment, identified drug abuse, retirement pension and ongoing pregnancy, patients lacking internet attached computers in their home.

Ethical considerations The Ethical application has been from the Regional Ethical Review Board in Umeå.

Procedure The study will be conducted in collaboration with a local physiotherapy unit in primary health care. We will actively recruit participants by advertising in local media.

Participants will be recruited through advertisements in local media. Each person answering the advert will get in contact with one of the researchers, who will give initial information of the study and then make an appointment for screening and assessment of whether the person is equivalent to the study's inclusion and exclusion criteria. Written information and written consent will be obtained for each participant included in the study.

Intervention The participants included in the study are randomized to one of two groups. The study begins with one group starting a baseline phase of 8 weeks where they are introduced into the web-based self-help program while the other group has a baseline phase of 6 weeks without any intervention. During the baseline phase, each participant answers a questionnaire with the outcome variables once /week. This is provided by the researchers.

The intervention consists of a web-based self-help program with cognitive behavioral therapy coaching in combination with individually tailored physiotherapy according to the person's needs for 16 weeks. All participants will receive an interactive web-based self-help pain program with coaching using CBT-principles individual coaching will be provided.One of the researchers will introduce each participant in the web-program. . A trained CBT-coach will be responsible for the coaching process during the intervention. The physiotherapy treatment is delivered at the physiotherapy unit, individualized for each patient, multimodal where treatment frequency and duration depends on the patient's needs. Initially in the intervention, each patient meets with the physiotherapist and the CBT-coach to synchronize the rehabilitation process according to the patient's needs and goals.

The web-based program The web-based program is based on CBT-principles, initially established by Livanda then further developed by Norrbotten County Council and Luleå University of Technology for a ongoing REHSAM II-project. The web-program consists of eight modules comprising; pain mechanism, activity balance and health, physical activity and ergonomics, emotions/ thoughts and behavior, stress and self-esteem, sleep, communication and conflicts, problem solving and planning future. The web-program includes informative texts, interactive media with questions for reflection and exercises to perform. As an example will each patient make their own activity plan and also reflect on priorities in life. The program also consists of instructional videos on for example ergonomics and relaxation exercises. The patient has the opportunities to play an active role in the web-program, as well as in the interaction with the CBT-coach. The aim of the program is to increase the patient's knowledge and understanding, supplying tools for coping in life-situation to increase health and work-ability.

The coaching process Within the program each participant formulates goals according to his/her individual pain rehabilitation needs in contact with the coach. The stepwise coaching process aims to fulfill each patient's individually formulated goals. The CBT-coach has a supportive role to guide the patient through the program and the rehabilitation using CBT-principles.

Outcome variables Primary outcome variables measured once a week during all the phases of the single subject experimental phase.

Self-perceived workability. This will be assessed by using the self-rated questionnaire Work Ability Index. By complementing outcome variables as Days of sick leave/activity compensation with Work Ability Index we will minimize the risk of a type II-error due to local labor market conditions.

Pain intensity. Average pain intensity during last 7 days in the musculoskeletal system will be measured by a Numeric Rating Scale (NRS).

Self-efficacy in relation to pain will be measured by Arthritis Self-efficacy scale (ASES:S); perceived capacity in relation to pain and perceived capacity in relation to other symptoms.

Considering the association of pain-related fear and self-reported occupational disability, kinesiophobia in relation to pain will be measured by the Swedish version of Tampa Scale of Kinesiophobia.

Health related quality of life. The Swedish version of RAND-36 will be used.

Also, the Patient Specific Functional Scale (PSFS) will be used to identify and measure activities rated important for each participant.

Analyses The design implies the study of a clinical progress in a controlled experimental manipulation by very frequent measurements of several outcome variables in a small sample of participants during a pre-intervention phase, an intervention phase and during an intervention withdrawal phase. 6 months after the intervention phase. The participants thereby act as their own controls and are seen as single systems in the analyses. The analyses focus on changes in levels, trends and variability in the outcome variables that can be attributed to the introduction of the intervention. Line graphs are used to describe the progress of the variables during the study phases for each of the participants, and visual analyses are enhanced by calculation of celeration lines and variability bands. The design cannot produce direct statistical inference, but it has the power to describe a clinical progress in detail in several individuals. Similarities between individuals will imply a certain transferability of results. The merits of this design as an additional tool to traditional group designs in the development of evidence based practice are described in a recent review.The design also allows for complementary analyses regarding for instance qualitative and quantitative data on the implementation of the intervention, experiences of the intervention from participants and therapists, costs, etc. This, together with analyses of outcome variables, can provide valuable knowledge regarding implementation in clinic.

Following the SSED design data will be analyzed on an individual level. For each participant, line graphs will display how outcome variables change along the measurement occasions throughout baseline and intervention phases. Analyses will be made as follows.

1. A visual analysis of whether changes in level and changes in slope of the outcome variable could be attributed to the introduction of the intervention. These analyses are complemented by the following calculations:
2. Calculation of +/-2SD bands for mean value of baseline phase. This is used in order to determine whether changes in level during (the later part of) the intervention phase could be seen as statistically significant when considering the variation during the baseline phase. This can be made either by determining if the mean value of the (later part of) the intervention phase is not within the +/- 2SD band, or by checking that at least 3 individual measurements in the intervention phase are outside the band.
3. Calculation of celeration lines. This is made to complement the analysis of change in trend (slope) of the outcome values throughout the phases. For each of the baseline and intervention phases, celeration lines are drawn between the median values for the first and second half of each phase and extended throughout the phase. The slopes of the lines are compared as to whether they differ substantially.

Complementary data Complementary data that will be collected within the project are activity logs from the web-based program (both participants and coach); number of coaching sessions and number of physiotherapy sessions. In addition, qualitative data from interviews with participants, coach and physiotherapists regarding e.g. experiences of process and results of the intervention will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Persons, with persistent or recurrent pain from the neck-shoulder or back, with a duration for at least three months,
* aged 18-63 years,
* scoring ≥ 90 on Linton´s questionnaire (indicating risk for continuous sick leave and development of persistent pain),
* who are disposable for labor market at least 25% are eligible for the study.
* They have to be fluent in the Swedish language.

Exclusion Criteria:

* Patients with dementia and/or restricted cognitive functioning.
* Persons with depression and/or anxiety. The latter will be screened with the Hospital Anxiety Depression Scale questionnaire.
* Terminally ill patients,
* comorbidity which might prevent treatment participation and ongoing causal treatment,
* identified drug abuse,
* retirement pension and ongoing pregnancy,
* patients lacking internet attached computers in their home.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Self-perceived workability. | Baseline, After intervention (16 weeks), 12 month
  Self-perceived workability. This will be assessed using the self-rated questionnaire Work Ability Index, which is a reliable and valid questionnaire addressing a persons perceived work capacity. By complementing outcome variables as Days of sick leave/activity compensation with Work Ability Index we will minimize the risk of a type II-error due to local labor market conditions.

SECONDARY OUTCOMES:
Health related quality of life | Baseline, After intervention (16 weeks), 12 month
  Health related quality of life will be measured using the RAND-36 questionnarie.

OTHER OUTCOMES:
Self-efficacy in relation to pain | Baseline, After intervention (16 weeks), 12 month
  Self-efficacy in relation to pain will be measured by Arthritis Self-efficacy scale (ASES:S); perceived capacity in relation to pain and perceived capacity in relation to other symptoms.
Pain intensity | Baseline, after intervention (16 weeks), 12 month
  Average pain intensity during last 7 days in the musculoskeletal system will be measured by a Numeric Rating Scale (NRS).

CONTACTS AND LOCATIONS:
Overall Officials: Mai Lindstrom, Dean, Principal Investigator — Luleå University of Technology
Locations (1):
- Luleå university of Technology, Luleå, Norrbotten County, Sweden